CLINICAL TRIAL: NCT07391592
Title: Post Market Clinical Follow-Up Study for EVOLUTION® NitrX™ Keeled Tibia and EVOLUTION® NitrX™ CS/CR Femur With Cruciate Sacrificing Insert
Acronym: NitrX
Status: Active, not recruiting | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 25DM0004
Record Dates: First submitted 2026-01-26; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthitis; Arthritis Knee; Joint Diseases; Avascular Necrosis; Rheumatoid Arthritis of Knee
MeSH Terms: conditions — Joint Diseases; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Newly or previously implanted patients: Single center, non-interventional prospective follow-up of newly or previously implanted subjects. Previously implanted subjects must be enrolled within 14 months of the study index surgery. Single study group with either newly or previously implanted patients with all EVOLUTION® NitrX™ components: Non-Porous Keeled Tibia, CS/CR Non-Porous Femur component, and EVOLUTION® MP CS tibial insert
  Interventions: Device: EVOLUTION® NitrX™

INTERVENTIONS:
Device: EVOLUTION® NitrX™ — EVOLUTION® NitrX™ Keeled Tibia and EVOLUTION® NitrX™ CS/CR Femur With Cruciate Sacrificing Insert

SUMMARY:
MicroPort Orthopedics Inc. (MPO) plans to market the EVOLUTION® NitrX™ Non-Porous Keeled Tibia and EVOLUTION® NitrX™ CS/CR Non-Porous Femur with the EVOLUTION® Cruciate Sacrificing (CS) Tibial Insert globally, including in the European Union (EU). MPO is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and effectiveness of the EVOLUTION® NitrX™ Non-Porous Keeled Tibia and EVOLUTION® NitrX™ CS/CR Non-Porous Femur. These components are used along with the EVOLUTION® Cruciate Sacrificing (CS) Tibial Insert components that is marketed in the European Union (EU). This type of data collection is required by regulatory authorities for all TKA devices that do not have medium to long-term clinical evidence available.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18 years of age at the time of surgery
* Subjects who were implanted with the Evolution® NitrX (SKU # listed below) in MicroPort Orthopedics' intended patient population listed within the Instructions for Use (IFU).
* Willing and able to participate in clinical study

Exclusion Criteria:

* Subjects without follow-up history
* Subjects not meeting the inclusion criteria
* Contraindications as listed in the IFU
* Currently enrolled in another study that could affect the endpoints of this protocol.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single study group with either newly or previously implanted patients with all Evolution® NitrX components: Non-Porous Keeled Tibia, CS/CR Non-Porous Femur component, and Evolution® MP CS Tibial insert.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score- Joint Replacement (KOOS JR) | 10 years
  KOOS is a validated patient-reported outcome measure designed to assess short- and long- term symptoms and functions in individuals with knee injuries and osteoarthritis. It is a 42-item questionnaire. KOOS JR is its short form, developed using Rasch analysis to provide a more efficient tool for clinical and research use. It has 7 items which measure pain, stiffness and function in daily life. Each item is scored from 0 (none) to 4 (extreme). The raw score (0-28) is converted to an interval score ranging from 0 to 100, where 100 indicates the best health and 0 means the worst health.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Sah, MD, Principal Investigator — Sah Orthopaedic Associates, Fremont, California, United States 94538
Locations (1):
- Sah Orthopaedic Associates, Fremont, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT07391592/Prot_000.pdf